CLINICAL TRIAL: NCT02189304
Title: A Phase I, Randomized, Double-Blind, Single-Dose, Three-Period, Three-Treatment, Cross-Over Study Evaluating the Pharmacokinetics and Safety of a Single Dose of PT010, a Single Dose of PT009, and a Single Dose of Open-Label Symbicort® Turbohaler® in Healthy Subjects
Brief Title: Pharmacokinetics and Safety Study of PT010 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT010002-00
Record Dates: First submitted 2014-07-09; First posted 2014-07-14 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: COPD
Keywords: Healthy volunteers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PT010 (Experimental): PT010; Budesonide, Glycopyrrolate, and Formoterol Fumarate Inhalation Aerosol. Administered as 2 inhalations
  Interventions: Drug: PT009; Drug: Symbicort Turbohaler
- PT009 (Experimental): PT009; Budesonide and Formoterol Fumarate Inhalation Aerosol. Administered as 2 inhalations
  Interventions: Drug: PT010; Drug: Symbicort Turbohaler
- Symbicort Turbohaler (Active Comparator): Symbicort Turbohaler; Budesonide and Formoterol Fumarate Inhalation Powder taken as 2 inhalations
  Interventions: Drug: PT010; Drug: PT009

INTERVENTIONS:
Drug: PT010 — PT010; Budesonide, Glycopyrrolate, and Formoterol Fumarate Inhalation Aerosol. Administered as 2 inhalations
  Other Names: PT010; Budesonide, Glycopyrrolate, and Formoterol Fumarate Inhalation Aerosol
  Arms: PT009; Symbicort Turbohaler
Drug: PT009 — PT009 administered as 2 inhalations
  Other Names: PT009; Budesonide and Formoterol Fumarate Inhalation Aerosol. Administered as 2 inhalations
  Arms: PT010; Symbicort Turbohaler
Drug: Symbicort Turbohaler — Symbicort Turbohaler taken as 2 inhalations
  Other Names: Symbicort Turbohaler; Budesonide and Formoterol Fumarate Inhalation Powder
  Arms: PT009; PT010

SUMMARY:
This is a single-center, Phase I, healthy adult subject study with a randomized, double blind, three period, three-treatment, cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form (ICF) prior to any study related procedures
* Male and female subjects 18 to 55 years, inclusive
* Good general health
* Medically acceptable contraception for women of child-bearing potential and males with female partners of childbearing potential
* Clinical labs within normal ranges or determined to be not clinically significant by the Investigator

Exclusion Criteria:

* Pregnancy, nursing female subjects, or subjects trying to conceive
* Clinically significant neurologic, cardiovascular, hepatic, renal, endocrinologic, pulmonary, hematological, psychiatric, or other medical illness that would interfere with participation in this study
* History of ECG abnormalities
* Cancer not in complete remission for at least 5 years
* Clinically significant, symptomatic prostatic hypertrophy
* Male subjects with a trans-urethral resection of the prostate or full resection of the prostate within 6 months prior to Screening
* Clinically significant bladder neck obstruction or urinary retention
* Inadequately treated glaucoma
* History of an allergic reaction or hypersensitivity to any drug or to any component of the formulations used in this study
* Subjects with pre-existing anemia and/or iron deficiency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2014-09-01 (Actual)

PRIMARY OUTCOMES:
Overall Safety of PT010, PT009 and Symbicort Turbohaler | 12 hours post dose
  The safety of PT010 and PT009 and Symbicort Turbohaler will be assessed based on physical examination, adverse events, vital signs, clinical laboratory values, and electrocardiogram

SECONDARY OUTCOMES:
◦Maximum plasma concentration (Cmax) of PT010, PT009 and Symbicort Turbohaler | 12 Hour post dose
◦Area under the curve from 0 to 12 hours (AUC0 12) of PT010, PT009 and Symbicort Turbohaler | 12 Hour post dose
◦Area under the curve from 0 to the time of the last measureable plasma concentration (AUC0 t) of PT010, PT009 and Symbicort Turbohaler | 12 Hour post dose
◦Area under the curve from 0 extrapolated to infinity (AUC0-∞) of PT010, PT009, and Symbicort Turbohaler | 12 Hour post dose
◦Time to maximum plasma concentration (tmax) of PT010, PT009, and Symbicort Turbohaler | 12 Hour post dose
◦Apparent terminal elimination half life (t½) of PT010, PT009, and Symbicort Turbohaler | 12 Hour post dose
◦Apparent total body clearance (CL/F) of PT010, PT009, and Symbicort Turbohaler | 12 Hour post dose
◦Apparent volume of distribution (Vd/F) of PT010, PT009, and Symbicort Turbohaler | 12 Hour post dose
◦Termination elimination rate constant (λz) of PT010, PT009, and Symbicort Turbohaler | 12 Hour post dose

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Orevillo, Study Chair — Pearl Therapeutics
Locations (1):
- SNBL Clinical Pharmacology Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Huang Y, Assam PN, Feng C, Su R, Dorinsky P, Gillen M. Ethnic pharmacokinetic comparison of budesonide/glycopyrrolate/formoterol fumarate metered dose inhaler (BGF MDI) between Asian and Western healthy subjects. Pulm Pharmacol Ther. 2020 Oct;64:101976. doi: 10.1016/j.pupt.2020.101976. Epub 2020 Nov 2. PMID 33152467
- [Derived] Maes A, DePetrillo P, Siddiqui S, Reisner C, Dorinsky P. Pharmacokinetics of Co-Suspension Delivery Technology Budesonide/Glycopyrronium/Formoterol Fumarate Dihydrate (BGF MDI) and Budesonide/Formoterol Fumarate Dihydrate (BFF MDI) Fixed-Dose Combinations Compared With an Active Control: A Phase 1, Randomized, Single-Dose, Crossover Study in Healthy Adults. Clin Pharmacol Drug Dev. 2019 Feb;8(2):223-233. doi: 10.1002/cpdd.585. Epub 2018 Jun 14. PMID 29901860